CLINICAL TRIAL: NCT01676623
Title: Impact Evaluation of a Social Franchise Model Implemented by Alive & Thrive for Improving Infant and Young Child Feeding and Child Nutrition in Rural Vietnam
Brief Title: Impact Evaluation of a Social Franchise Model for Improving Infant and Young Child Feeding and Child Nutrition in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IFPRI-S-01 (2)
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Child Nutrition; Stunting; Exclusive Breastfeeding; Complementary Feeding
Keywords: Child nutrition; Stunting; Exclusive breastfeeding; Complementary feeding; Social franchise; Mass media; Counseling; Facility-based
MeSH Terms: conditions — Growth Disorders; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison area, only standard government services (Active Comparator): This intervention arm will receive the standard government services offered at CHCs all over Vietnam. In addition, participants in this arm will be exposed to the nationwide mass media campaign.
  Interventions: Behavioral: Standard government health services; Behavioral: Mass media campaign
- A&T Franchise (Experimental): In this arm, the 20 CHCs will offer Alive & Thrive branded franchise services with enhanced quality of IYCF counseling through interpersonal contact between health workers at the commune level and clients who use the commune health services. In addition, the clients could also be exposed to the mass media campaign.
  Interventions: Behavioral: Standard government health services; Behavioral: Alive & Thrive IYCF franchise services; Behavioral: Mass media campaign

INTERVENTIONS:
Behavioral: Standard government health services — This intervention will be basic preventive and curative health services provided by the commune health centers. This includes antenatal care, postnatal care and basic nutrition related counseling.
Behavioral: Alive & Thrive IYCF franchise services — This intervention includes intensive behavioral counseling to improve infant and young child feeding. A package of 15 counseling contacts that are quality assured and branded will be offered to families of infants and young children. Services might also include user fees.
  Arms: A&T Franchise
Behavioral: Mass media campaign — Alive & Thrive is implementing a nationwide mass media campaign in 2011, 2012 and 2013, with a focus on improving breastfeeding practices. The mass media intervention includes TV and radio spots as well as an internet site and a telephone hotline.

SUMMARY:
Alive & Thrive is an initiative that aims to improve infant and young child feeding practices and reduce childhood stunting. In Vietnam, Alive & Thrive's primary intervention is implemented through a social franchise linked with the government's health system. The impact evaluation is conducted using a cluster-randomized design in which 20 commune health centers (CHC) were assigned to the social franchise model, and 20 CHC were assigned to routine government services. Repeated cross-sectional baseline and endline surveys will be used to assess the public health impact of this intervention. The baseline was in 2010 and an endline survey in the same communities will be conducted in 2014. Mixed methods process evaluation will be conducted in 2011, 2012 and 2013 to study the pathways through which the program impact is achieved.

DETAILED DESCRIPTION:
Link provided to journal manuscript describing design of evaluation provides additional detail: http://fnb.sagepub.com/content/34/3_suppl2/S195.full.pdf

ELIGIBILITY:
Inclusion Criteria:

* Children 0-60 months of age

Exclusion Criteria:

* None

Max Age: 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4000 (Actual)
Dates: Start 2010-04; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding among children 0-6 months of age | 4 years
  Exclusive breastfeeding in children 0-6 months of age is one of the eight WHO-recommended IYCF core indicators will be measured to capture breastfeeding and complementary feeding practices. It is measured using survey based recall by interviewing mothers of children in the age group for the indicator.
Child heights and weights (children 24-60 months of age) | 4 years
  Heights and weights of children in the intervention and comparison communes covered by the CHCs in the study will be assessed in 2014. A new sample of children 24-60 months will be measured in the repeated cross-sectional endline survey to measure these outcomes and compute height-for-age, weight-for-age and weight-for-height z-scores based on the WHO growth reference standards.
Complementary feeding for children 6-23.9 months of age | 4 years
  Indicators of complementary feeding - diet diversity, minimum acceptable diet, and minimum meal frequency, measured in children 6-23.9 months of age are one of the eight WHO-recommended IYCF core indicators will be measured to capture breastfeeding and complementary feeding practices. These are measured using survey based recall by interviewing mothers of children in the age group for the indicator.

SECONDARY OUTCOMES:
Early initiation of breastfeeding in children 0-24 months of age | 4 years
  Early initiation of breastfeeding (in the first hour after birth) is measured in children 0-23.9 months of age and it is one of the eight WHO-recommended IYCF core indicators will be measured to capture breastfeeding and complementary feeding practices. These are measured using survey based recall by interviewing mothers of children in the age group for the indicator. Samples for children 0-6 months and 6-23.9 are combined to calculate this indicator

CONTACTS AND LOCATIONS:
Overall Officials: Purnima Menon, PhD, Principal Investigator — International Food Policy Research Institute; Rahul Rawat, PhD, Principal Investigator — International Food Policy Research Institute; Phuong Nguyen, PhD, Principal Investigator — International Food Policy Research Institute; Marie T Ruel, PhD, Principal Investigator — International Food Policy Research Institute
Locations (1):
- Alive & Thrive & International Food Policy Research Institute, Hanoi, Hanoi, Vietnam

REFERENCES:
- [Derived] Kim SS, Nguyen PH, Tran LM, Alayon S, Menon P, Frongillo EA. Different Combinations of Behavior Change Interventions and Frequencies of Interpersonal Contacts Are Associated with Infant and Young Child Feeding Practices in Bangladesh, Ethiopia, and Vietnam. Curr Dev Nutr. 2019 Dec 9;4(2):nzz140. doi: 10.1093/cdn/nzz140. eCollection 2020 Feb. PMID 31976385
- [Derived] Nguyen PH, Kim SS, Tran LM, Menon P, Frongillo EA. Intervention Design Elements Are Associated with Frontline Health Workers' Performance to Deliver Infant and Young Child Nutrition Services in Bangladesh and Vietnam. Curr Dev Nutr. 2019 Jul 10;3(8):nzz070. doi: 10.1093/cdn/nzz070. eCollection 2019 Aug. PMID 31346584
- [Derived] Rawat R, Nguyen PH, Tran LM, Hajeebhoy N, Nguyen HV, Baker J, Frongillo EA, Ruel MT, Menon P. Social Franchising and a Nationwide Mass Media Campaign Increased the Prevalence of Adequate Complementary Feeding in Vietnam: A Cluster-Randomized Program Evaluation. J Nutr. 2017 Apr;147(4):670-679. doi: 10.3945/jn.116.243907. Epub 2017 Feb 8. PMID 28179488
- [Derived] Menon P, Nguyen PH, Saha KK, Khaled A, Kennedy A, Tran LM, Sanghvi T, Hajeebhoy N, Baker J, Alayon S, Afsana K, Haque R, Frongillo EA, Ruel MT, Rawat R. Impacts on Breastfeeding Practices of At-Scale Strategies That Combine Intensive Interpersonal Counseling, Mass Media, and Community Mobilization: Results of Cluster-Randomized Program Evaluations in Bangladesh and Viet Nam. PLoS Med. 2016 Oct 25;13(10):e1002159. doi: 10.1371/journal.pmed.1002159. eCollection 2016 Oct. PMID 27780198
- See also: Alive & Thrive's overall web page. Includes description of Vietnam program. — http://www.aliveandthrive.org